CLINICAL TRIAL: NCT03508895
Title: Double-blind, Randomized, Cross-over Trial of Whole Hemp Seed Protein and Hemp Seed Protein Hydrolysate Derived Bioactive Peptide Consumption for Hypertension
Brief Title: Hemp Seed Protein and Bioactive Peptides Consumption for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Manitoba Harvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HS20390 (B2016:125)
Record Dates: First submitted 2018-03-29; First posted 2018-04-26 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Hemp seed protein; Protein hydrolysate; Bioactive peptides; Cannabis sativa; High blood pressure
MeSH Terms: conditions — Hypertension; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole hemp seed protein (Experimental): 25 grams of hemp seed protein powder, twice a day
  Interventions: Other: Whole hemp seed protein
- Whole hemp seed protein plus bioactive peptides (Experimental): 22.5 grams of hemp seed protein and 2.5 grams of hemp seed protein hydrolysate derived bioactive peptides, twice a day
  Interventions: Other: Whole hemp seed protein plus bioactive peptides
- Casein protein (Active Comparator): 25 grams of protein powder, twice a day
  Interventions: Other: Casein protein

INTERVENTIONS:
Other: Whole hemp seed protein — The intervention was provided in the form of a smoothie.
  Arms: Whole hemp seed protein
Other: Whole hemp seed protein plus bioactive peptides — The intervention was provided in the form of a smoothie.
  Arms: Whole hemp seed protein plus bioactive peptides
Other: Casein protein — The intervention was provided in the form of a smoothie.
  Arms: Casein protein

SUMMARY:
This clinical trial is being conducted to study the effect of whole hemp seed protein, hemp seed protein hydrolysate derived bioactive peptide and casein protein consumption on systolic and diastolic ambulatory blood pressure. This study is will be conducted in 35 hypertensive participants aged between ≥18 and ≤75 yrs who have systolic blood pressure higher than 130 mmHg or diastolic blood pressure ≤ 110 mmHg. The study will consist of 3 periods of 42 days each during which participants will consume assigned treatment. Consumption of treatments will be from days 1 to 42. There will also be a washout period of a minimum of 14 days between the 3 treatment periods where the participants can consume their habitual diets. The entire study is designed to take 22 weeks from start to completion. The participants will consume the assigned treatment twice a day. The treatments are in the form of a smoothie and the smoothies will consist of frozen fruit, fruit juice, frozen yoghurt/sorbet, and 25 g of protein from treatment protein powder which is 25 grams of casein protein, 25 grams of hemp seed protein, or 22.5 grams of hemp seed protein and 2.5 grams of hemp seed protein hydrolysate derived bioactive peptides. On days 1 and 42 of each treatment period of the trial, body weight, waist and hip circumference, blood pressure, pulse wave velocity (PWV) and augmentation index (AI) will be measured. Ambulatory blood pressure (ABP) over 24 hours will also be measured on day 1 of phase 1 and day 42 of each treatment period of the trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-40 kg/m2
* Systolic blood pressure between 130-160 mmHg
* Diastolic blood pressure ≤ 110 mmHg
* Ability and willingness to give informed consent to participate in the trial
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
* Willingness to fast 10-12 hours before blood samples and abstain from alcohol two days prior to blood sampling and BP measurement and abstain from coffee and physical exercise at least 14 and 4 hours before measurement respectively
* Negative pregnancy test for women with child-bearing potential

Exclusion Criteria:

* Unable to speak/read in English
* Active cardiovascular disease including stroke, congestive heart failure, myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, temporal ischemic attacks, secondary hypertension, type 1 or type 2 diabetes, anemia, abnormal electrolytes, proteinuria, and abnormal liver, kidney or thyroid function
* History of cancer or malignancy in the last 5 years, or any metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which could interfere with the results of the study or the safety of the participant
* Taking lipid or blood pressure lowering medications or any type of supplements for less than 3 months (Note: all medications or supplements will be permitted if they are on a stable dose for more than 3 months before the start of the study)
* Smokers, tobacco/snuff/nicotine users, recreational drug users
* Consuming more than 14 alcoholic beverages a week
* Any dietary restrictions preventing from consuming the trial treatments
* Weight gain or loss greater than 5 kg in the past three months
* Exercising > 15 miles/wk or 4,000 kcal/wk
* Known to be pregnant or breast-feeding or planning on becoming pregnant during the trial period
* Having clinically significant biochemistry defined as: Sodium: <134 mmol/l, >148 mmol/l; fasting glucose: > 6.1 mmol/L; LDL-C ≥4.9 mmol/L or any other clinically significant abnormality in hematology and/or biochemistry at the investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour ambulatory blood pressure | Measured at day 1 of phase 1 (baseline) and change from baseline ABP at week 6 of phase 1, 2 and 3
  Participants were fitted with an ambulatory blood pressure monitor (ABPM) for 24 hours. Continuous diastolic and systolic blood pressure were measured over 24 hours.

SECONDARY OUTCOMES:
Change in serum renin concentration | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline serum renin concentration at day 42 of phase 1, 2 and 3
  Measured using a fluorometric microplate reader (Spectra MAX Gemini, Molecular Devices, Sunnyvale, CA).
Change in angiotensin-converting enzyme (ACE) activity in the plasma | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline plasma ACE activity at day 42 of phase 1, 2 and 3
  Measured using spectrophotometric method with furanacryloyl-L-phenylalanylglycylglycine (FAPGG) as substrate
Change in nitric oxide (NO) plasma concentrations | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline plasma NO concentration at day 42 of phase 1, 2 and 3
  Was determined in plasma using nitrate/nitrite colorimetric assay kit (Cayman Chemical, Michigan, USA)
Change in plasma reactive oxygen and nitrogen species (ROS/RNS) concentration | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline ROS/RNS concentration at day 42 of phase 1, 2 and 3
  Was determined using OxiSelec ROS/RNS assay kit and fluorescence plate reader at 480 nm excitation / 530 nm emission
Change in plasma total peroxides (PTPs) concentration | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline PTPs concentration at day 42 of phase 1, 2 and 3
  Was determined using microplate reader at 500 nm
Change in plasma superoxide dismutase (SOD) concentration | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline plasma SOD concentration at day 42 of phase 1, 2 and 3
  SOD OxiSelect assay kit (Cell Biolabs, Inc., San Diego, CA, USA) and microplate reader at 490 nm were used for this assay
Change in plasma catalase (CAT) concentration | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline plasma CAT concentration at day 42 of phase 1, 2 and 3
  CAT assay kit (Cell Biolabs, Inc. San Diego, CA, USA) and fluorescence microplate reader at excitation and emission 550 and 590 nm were used for this assay
Change in plasma free oxylipin concentrations | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline plasma free oxylipin concentrations at day 42 of phase 1, 2 and 3
  HPLC/MS/MS by using a Luna 5μm C18 column on a Shimadzu Nexera XR HPLC, coupled to an ABSciex QTRAP 6500 MS

OTHER OUTCOMES:
Change in blood pressure | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline blood pressure at week 3 and 6 of phase 1, 2 and 3
  Systolic and diastolic blood pressure were measured using an automated oscillometric measurement device in an office setting in a quiet room while the participant wass in a seated position and arm rested on an arm rest at heart level. Participants were advised to rest quietly throughout the measurements. Measurements were performed 4 times at 2-minute intervals.
Change in pulse wave velocity (PWV) | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline PWV at week 6 of phase 1, 2 and 3
  Measured using an automated oscillometric measurement device (Mobil-O-Graph, IEM, Stolberg, Germany) in an office setting in a quiet room while the participant was in a seated position and arm rested on an arm rest at heart level. Participants were advised to rest quietly throughout the measurements.
Change in augmentation index (AI) | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline AI at week 6 of phase 1, 2 and 3
  Measured using an automated oscillometric measurement device (Mobil-O-Graph, IEM, Stolberg, Germany) in an office setting in a quiet room while the participant was in a seated position and arm rested on an arm rest at heart level. Participants were advised to rest quietly throughout the measurements.
Change in body weight | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline body weight at week 6 of phase 1, 2 and 3
  Following standardized procedures
Change in waist circumference | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline waist circumference at week 6 of phase 1, 2 and 3
  Following standardized procedures
Change in hip circumference | Measured at day 1 of phase 1, 2 and 3 (baseline) and change from baseline hip circumference at week 6 of phase 1, 2 and 3
  Following standardized procedures
Change in body composition | Measured at day 1 of phase 1 (baseline) and change from baseline body composition at week 6 of phase 1, 2 and 3
  Looking at potential changes in body fat and lean mass composition by Dual X-ray absorptiometry (DXA). For this procedure, the participant were needed to lie in a horizontal position for about 5-15 minutes while the scan arm passes from the head to the feet. The radiation from this test was very low dosage (equivalent to approximately 1 day of natural background radiation).

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi Aluko, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Food Technology and Research, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Samsamikor M, Mackay DS, Mollard RC, Alashi AM, Aluko RE. Hemp seed protein and its hydrolysate compared with casein protein consumption in adults with hypertension: a double-blind crossover study. Am J Clin Nutr. 2024 Jul;120(1):56-65. doi: 10.1016/j.ajcnut.2024.05.001. Epub 2024 May 4. PMID 38710445
- [Derived] Samsamikor M, Mackay D, Mollard RC, Aluko RE. A double-blind, randomized, crossover trial protocol of whole hemp seed protein and hemp seed protein hydrolysate consumption for hypertension. Trials. 2020 Apr 23;21(1):354. doi: 10.1186/s13063-020-4164-z. PMID 32326966